CLINICAL TRIAL: NCT02712957
Title: A Proof-of-Concept, Randomized, Double Blind, Placebo and Active Control, 3-Period, Crossover Design Study Assessing NEO6860 in Patients With Pain Associated With Osteoarthritis of the Knee
Brief Title: A Proof-of-Concept Study Assessing NEO6860 in Osteoarthritis Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neomed Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NEO6860-OA-01
Record Dates: First submitted 2016-03-09; First posted 2016-03-18 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Pain; Osteoarthritis of the Knee
MeSH Terms: conditions — Pain; Osteoarthritis, Knee | interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- NEO6860 (Experimental): NEO6860 is provided as a powder in individual containers to be reconstituted as a suspension. In this arm patients will receive both NEO6860 and a placebo of naproxen.
  Interventions: Drug: NEO6860; Drug: Naproxen placebo
- Placebo (Placebo Comparator): In this arm, patients will receive both placebo: oral liquid suspension (NEO6860 placebo) and capsule (naproxen placebo).
  Interventions: Drug: NEO6860 placebo; Drug: Naproxen placebo
- Naproxen (Active Comparator): Naproxen is provided as over-encapsulated tablets using a commercially approved medication. In this arm patients will receive both naproxen and a placebo of NEO6860.
  Interventions: Drug: NEO6860 placebo; Drug: Naproxen

INTERVENTIONS:
Drug: NEO6860 — TRPV1 antagonist
  Arms: NEO6860
Drug: NEO6860 placebo — Inactive substance
  Arms: Naproxen; Placebo
Drug: Naproxen — NSAID
  Arms: Naproxen
Drug: Naproxen placebo — inactive substance
  Arms: NEO6860; Placebo

SUMMARY:
The purpose of this study is to assess NEO6860, a modality selective TRPV1 antagonist, in patients with pain associated with osteoarthritis of the knee.

DETAILED DESCRIPTION:
The study will be randomized, double blind, placebo and active control, a 3-way, 3-period crossover design, where each of the estimated 50 enrolled patients will receive alternately (i) NEO6860 (500 mg bid), (ii) placebo and (iii) Naproxen (500 mg bid). To ensure blinding, double dummy techniques will be used, so that at each period, patient will receive an oral liquid suspension (NEO6860 or its placebo) and one capsule (naproxen or its placebo).

Following a screening period, a maximum of 28 days before dosing, subjects will be randomized to one of the scheduled sequences. At each dosing period, subjects will be requested to participate in 2 clinic visits:

* One residential visit, the morning of investigational product dosing. Subjects will stay in the Clinical Research Unit approximately 13 hours
* One end of period visit, 24 h after first dosing A total of 2 washout periods of 1 to 3 weeks will separate the dosing periods. Once the 3 dosing periods will be completed, the subjects will come back to the clinic for a follow up visit (7 to 10 days post last dose).

Note: for a subpopulation, at one site, an assessment of heat pain threshold and tolerance will be conducted requiring a residential period of approximately 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.0 and 35.0 kg/m2 inclusive;
* Patients diagnosed with osteoarthritis of the knee, according to American College of Rheumatology (ACR) guidelines, by meeting at least 3 of the following: age > 50, morning stiffness < 30 minutes, crepitus on active motion, bone tenderness, bone enlargement, no palpable warmth of synovium;
* Grade I, II or III using Kellgren-Lawrence classification on an X-Ray of the knee
* WOMAC pain subscale ≥ 8
* R square of the Focused Analgesia Selection Task (FAST) outcome value greater than 0.70

Exclusion Criteria:

* Patients with, or with a history of, any clinically significant disorders (including fibromyalgia and other painful disorders) which may interfere with the primary objectives of the study
* Patients treated in the previous 3 months with topical capsaicin or intra-articular corticosteroids;
* Patients with a contra-indication for the use of Naproxen or acetaminophen;

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-03; Primary Completion 2016-11-17 (Actual); Study Completion 2016-11-24 (Actual)

PRIMARY OUTCOMES:
Mean change in Numerical Rating Scale (NRS, 0-10) from baseline after the staircase test to 8 hours post first dose after the staircase test on the index knee. | 8 hours post dosing. This endpoint will be collected 3 times, 8 hours post dosing for each period: NEO6860, naproxen and placebo.
  Patients are asked to step fully up onto a 8-inch (20 cm) high platform with both feet and back down a total of 24 times.

SECONDARY OUTCOMES:
WOMAC 3.1 Index Likert pain subscale | from baseline (screening) to 24 hour recall post 1 day treatment at each of the 3 periods
Patient's Global Impression of Change (PGIC) | 24 hour post 1 day treatment at each of the 3 periods

CONTACTS AND LOCATIONS:
Overall Officials: Dan A Chiche, MD, Study Director — Neomed Institute
Locations (3):
- Canada (3):
  - Diex Recherche Montreal Inc, Montreal, Quebec
  - Algorithme Pharma, Montreal, Quebec
  - Diex Recherche Sherbrooke Inc, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No